CLINICAL TRIAL: NCT01020513
Title: Subcutaneous Recombinant Human Hyaluronidase: Workflow Analysis and Emergency Department Design
Acronym: Hylenex-ED
Status: Withdrawn | Type: Observational
Why Stopped: This study was closed before accrual due to FDA recall of Medication
Sponsor: University of California, San Diego (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, John Fontanesi, Professor, University of California, San Diego
Other Study IDs: UCSD-2010-0250
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study examining the workflow dynamics and training requirements that support effective use of subcutaneous hydration delivery (a newly FDA approved Baxter product) compared to standard intravenous hydration/medication delivery. Emergency departments already using both Subcutaneous Recombinant Human Hyaluronidase and standard IV hydration will be enrolled. Patients will be receiving the hydration method selected by their emergency department physician and the investigators will then observe:

1. Patient Throughput

   * Efficiency of patient care and treatment areas
   * Safety of patient care and treatment areas
   * Support Service processes that impact patient flow
2. Clinical Outcomes

   * Time to conversion from dehydration to hydration'
   * Rate of complications
3. Satisfaction

   * Staff satisfaction with Subcutaneous hydration vs. Intravenous hydration
   * Patient satisfaction with Subcutaneous hydration vs. Intravenous hydration

DETAILED DESCRIPTION:
SPECIFIC AIMS This study examines the operational consequences and training requirements for implementing subcutaneous hydration vs. standard intravenous hydration in emergency departments.

B. BACKGROUND AND SIGNIFICANCE Emergency departments across the nation are overcrowded. Emergency department visits hit a new high in 2005, with more than 115 million visits, an increase of 5 million visits over the previous year, and a 20 percent increase over 10 years. During the same period the number of hospital EDs decreased more than 9 percent from 4,176 to 3,795. A consequence of the increase in demand occurring during a decrease in capacity, according to the American College of Emergency Physicians is that 60 percent of EDs report that the overcrowding has forced their facilities to divert patients and though more than 70 percent of hospitals reported having a goal of admitting patients within two hours of arrival in the emergency department, almost half of that group routinely fails.

Overcrowding not only results in delayed treatment, long patient waiting time, overburdened working staff, patient elopement, and low throughput, it also results in increased medical errors due to overloading and significant legal and financial risks.

These issues have led to a number of initiatives with, potentially the most profound being the 2007 Joint Commission requirement ( Leadership Standard, LD.3.15) requiring hospital leadership to:"… develop and implement plans to identify and mitigate impediments to efficient patient flow throughout the hospital".

Developing processes and procedures that can improve patient ﬂow in EDs, improve efficiency and reduce crowding is in all parties interests.

One potential area of improvement is in the hydration of patients. Twenty-five million Americans have intravenous catheters placed each year representing significant commitment of time, personnel, and resources. Several systems have been devised for the effective delivery of injectable material into a body using intravenous systems, but all suffer from drawbacks including trauma associated with intravenous needle placement and swelling, infection and limited, often compromised, placement sites . Furthermore intravenous hydration delivery require, at minimum, an RN who not only starts the IV but is also expected to monitor rates of perfusion (Adequate end-organ perfusion is best indicated by urine output of > 0.5 to 1 mL/kg/h) and notify the physician when desired end-states are obtained. In our own studies of Emergency Departments, this process added significant time to patient stays as well as increased error rates in the form of either ration fluids running out without replacement or patients needing to urinate without a Nurse recording that they had reached this end-point.

Improvement in either the rate of hydration and reduction in trauma and complications associated with typical intravenous systems should be a benefit to both patients and health care systems. Healthcare has developed a new system of hydration/medication delivery using Subcutaneous Recombinant Human Hyaluronidase. Subcutaneous Recombinant Human Hyaluronidase offers several advantages in hydrating emergency department patients over I.V. hydration methods. These include unlimited placement sites, (providing both psychological and physiological benefits), more rapid hydration, potentially administered by lower-cost and more available ED personnel than required for IVs.

However, new technologies super-imposed on old processes frequently do not generate the full potential of the new technology. Cars required a paved highway system and cell-phones required methods for uniquely identifying individual calls in three dimensional space. Attempting to implement Subcutaneous Hydration in an environment such as an Emergency Department may find "as is" workflow dynamics and skills do not effectively support the new technology. It is essential to understand how Emergency rooms function to understand how to improve the process, and where training in use of new technologies is most appropriately addressed to realize efficiencies and improved quality of care. Following is our model of EDs:

D. RESEARCH DESIGN AND METHODS This is a classic direct observation, workflow study in which the endpoints are the (potential) time differences in patient throughput, when hydration occurs via Subcutaneous Recombinant Human Hyaluronidase vs. Intravenous methods. We will also capture difference in patient and staff satisfaction for the two hydration methods. The satisfaction survey occurs immediately as part of the workflow observation.

The study design employs a Difference within Difference design in which the relative differences in patient throughput (primary variable of interest) and patient/staff satisfaction (secondary variable of interest for the various hydration/medication delivery systems is assessed at each site. It is the relative difference in measures for each site that is used in the aggregate for analysis. This mitigates the danger of large variations between sites overwhelming the differences between treatment options within sites.

Since this is an observational study, primarily of workflow characteristics, we will not (nor could we) make any determination of the appropriateness of individual provider's decision to either initiate or discontinue patient hydration.

Approach Between three and five Emergency Departments (depending on volume) that have already approved Subcutaneous Recombinant Human Hyaluronidase for their formulary will be included in this study. Following UCSD (and other relevant participating organizations) IRB approval, the UCSD P.I. and Project Coordinator will coordinate with identified administrative personnel at each research site regarding the nature of the study, provide an introduction of field observers, and what the product of the study will be. In addition, each site will be asked if there are specific issues they would like the research team to analyze that fit within the parameters of the study. Once all clearances and permissions are obtained, field observers will be oriented to the individual facilities and introduced to the staff.

Observations will be conducted in the following manner, field staff will observe ED patients and record the time they enter the facility. Once ED patients have completed the triage and are identified as an Acuity Level 3-5, field staff will approach ED patients and offer the opportunity to participate in the observational study. If signed permission is granted then field staff will "shadow" patients through the total ED visit using the Observational Checklist of Patient Encounters (OCPE), which has been published by the Joint Commission. 15 It is a 52 item checklist capturing three types of data:

1. Operational conditions at the time of an encounter (e.g. staffing ratios X number of patients)
2. Whether key procedures occurred (e.g. temperature taken, pain assessment completed)
3. Time to task completion (e.g. how long from the time an imaging study was ordered until the patient is taken to imaging) Patient satisfaction data will be collected as part of each workflow observation. Secondary variables of interest, specifically satisfaction and assessment of possible iatrogenic effects, occur at the conclusion of each observation. Patients are directly surveyed about their satisfaction with the encounter. Preference items (e.g. satisfaction with the provider) use standard 5-point likert scale while objective items (e.g. "is the care you received the care you expected, did you have any bruising around the hydration site) are cast as binary answers. Staff and providers undergo similar direct surveys of satisfaction and observation of iatrogenic effects, though the interview is not time-dependent as the patient satisfaction surveys.

Outcome Measures The data generated by the workflow observations and satisfaction surveys produce three distinct types of data sets for analysis. The one of primary interest for this study is the difference in time sequences and patient throughput between Subcutaneous Recombinant Human Hyaluronidase vs. Intravenous hydration methods. This type of data not only provides simple time-motion comparisons, it is also frequently used to generate measures of efficiency (i.e. how many patients can be hydrated for a given unit of time and labor) and proficiency (i.e. how many patients can be correctly hydrated for a given unit of time and labor). Secondary outcomes of interest include the difference in patient and staff satisfaction, including perception of iatrogenic effects, between Subcutaneous Recombinant Human Hyaluronidase and Intravenous hydration methods. The third data set includes the operational conditions requisite for effective use of Subcutaneous Recombinant Human Hyaluronidase use.

Data Analysis Data preparation and analysis will follow standard statistical techniques appropriate for each method used in this study. For example, McNemar tests will be used to determine significant changes for dichotomous variables such as errors of commission and omission (e.g., IV fluid ran out, patient urinates without staff noting). Paired-samples t-tests will be used to determine significant differences for both discrete continuous variables (e.g., time required to perform exam, time in waiting room) and ratio variables (e.g., patient/provider time to all time in clinic, patient/provider time to waiting time in the exam room). Wilcoxon signed-rank tests will be used to determine significant changes for variables using Likert scale response options (e.g., provider, staff, and patient satisfaction ratings on a 5-point scale).

Outcome measures of efficiency, such as improved patient throughput or increased adherence to ED policy and procedures, will use traditional parametric efficiency calculations. Efficiency is essentially how much of a service can be provided correctly for a given unit of time and resources (including personnel). Efficiency will be calculated using the following formula:

Where:

N = individuals who could be hydrated PV = probability of being hydrated with Subcutaneous Recombinant Human Hyaluronidase PHHR = probability of hydration that has begun evaluated within time defined by protocol PD = probability of hydration iatrogenic effects L = labor costs C = capital costs M = material costs

Finally, data will undergo Critical Path Analysis to identifying "inputs" or operational factors controlling patient flow dynamics and clinical outcomes. This analysis will use classification and regression analysis using binary recursive partitioning to identify the variables with the greatest predictive ability to correctly classify patient's lengths of stay in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Triaged as stage 3 or more (less acute)

Exclusion Criteria:

* Triaged as stage 2 or less (more acute), AND arriving for purposes of forensic/criminal evaluations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: non-emergent patients in Emergency Departments
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
elapsed time in Emergency Department | elapsed time in the Emergency Department is measured from the point a patient enters until they leave
  it is hypothesized patients hydrated via Subcutaneous Recombinant Human Hyaluronidase will progress to discharge from the emergency department faster then will patients hydrated via I.V.

CONTACTS AND LOCATIONS:
Overall Officials: John M Fontanesi, PhD, Principal Investigator — UCSD School of Medicine, Department of General Internal Medicine